CLINICAL TRIAL: NCT00745654
Title: Chronic Pain After Lung Transplantation, an Incidence Study
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: MD, Kim Wildgaard, Section for Surgical Pathophysiology 4074
Other Study IDs: H-B-2008-058; 2007-58-0015
Record Dates: First submitted 2008-07-30; First posted 2008-09-03 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-09

CONDITIONS: Lung Transplantation
Keywords: Lung Transplantation; Chronic pain; Thoracotomy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an investigation on the frequency of chronic pain amongst recipients after lung transplantation. Factors relating to the development of chronic pain are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give consent
* Can read
* Residing in Denmark

Exclusion Criteria:

* Unable to understand the written information in Danish
* Abuse (Medicine, Drugs, Alcohol)
* Severe psychiatric Illness
* Conflicting neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post lung transplantation patients in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Wildgaard, MD, Principal Investigator — Section for Surgical Pathophysiology 4074; Henrik Kehlet, MD,Phd,Proff, Study Chair — Section for Surgical Pathophysiology 4074
Locations (1):
- Section for Surgical Pathophysiology 4074, Copenhagen, Denmark